CLINICAL TRIAL: NCT06871410
Title: CD83 CAR T in Relapsed or Refractory Acute Myeloid Leukemia (AML): A Phase I Trial
Brief Title: Genetically Engineered Cells (CD83 CAR T Cells) for the Treatment of Relapsed or Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-3916824; NCI-2025-01523 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-3916824 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2025-03-10; First posted 2025-03-12 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Specimen Handling; X-Rays; Cyclophosphamide; fludarabine phosphate; Hydroxyurea; Leukapheresis; Spinal Puncture; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (fludarabine, cyclophosphamide, CD83 CAR T-cells) (Experimental): Patients undergo leukapheresis to obtain PBMCs for CD83 CAR T-cell product manufacturing on day -21 and may receive hydroxyurea at the discretion of the treating physician on study. Patients then receive fludarabine IV over 30 minutes and cyclophosphamide IV over 2 hours on days -5 to -3 in the absence of disease progression or unacceptable toxicity. Patients then receive CD83 CAR T-cells IV over 15 minutes on day 0. Patients also undergo ECHO and chest x-ray during screening, blood sample collection throughout the study, and CT and/or PET, as well as lumbar puncture as clinically indicated. In addition, patients may undergo bone marrow aspiration throughout the study.
  Interventions: Drug: Autologous Anti-CD83 CAR T-cells; Procedure: Biospecimen Collection; Procedure: Chest Radiography; Procedure: Computed Tomography; Drug: Cyclophosphamide; Procedure: Echocardiography; Drug: Fludarabine Phosphate; Drug: Hydroxyurea; Procedure: Leukapheresis; Procedure: Lumbar Puncture; Procedure: Positron Emission Tomography; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Autologous Anti-CD83 CAR T-cells — Given IV
  Other Names: Autologous Anti-CD83 CAR T Cells; Autologous Anti-CD83 CAR-T Cells
Procedure: Biospecimen Collection — Undergo bone marrow aspiration blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Chest Radiography — Undergo chest x-ray
  Other Names: Chest X-ray
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Drug: Hydroxyurea — Given hydroxyurea
  Other Names: Droxia; Hydrea; Hydroxycarbamide; Litalir; Onco-Carbide; Oncocarbide; Oxeron; SQ 1089; SQ-1089; Syrea; WR 83799
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocyte Adsorptive Apheresis; Leukocytopheresis; Therapeutic Leukopheresis; White Blood Cell Reduction Apheresis
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of genetically engineered cells (CD83 chimeric antigen receptor [CAR] T cells) in treating patients with acute myeloid leukemia (AML) that has come back after a period of improvement (relapsed) or has not responded to previous treatment (refractory). CD83 is a protein that is found on AML blasts. Blasts are abnormal immature white blood cells that can multiply uncontrollably: filling up the bone marrow and preventing the production of other cells important for survival. CD83 CAR T cells represent a new cell therapy to eliminate AML blasts, while avoiding the risk for graft versus host disease (GVHD) after stem cell transplant to replace bone marrow or, tumor toxicity like myeloid aplasia where the body's own immune system causes damage to the bone marrow stem cells. Therefore, human CD83 CAR T cells are a promising cell-based approach to preventing two critical complications of stem-cell transplant - GVHD and relapse. Giving CD83 CAR T cells may be safe, tolerable, and/or effective in treating patients with relapsed or refractory AML.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and determine the maximal tolerated dose (MTD) of autologous anti-CD83 CAR T-cells (CD83 CAR T cells) administered as a single infusion to refractory/relapsed acute myeloid leukemia (AML) patients.

SECONDARY OBJECTIVES:

I. To observe and record activity against AML. II. To evaluate response for AML using 2022 European Leukemia Net (ELN) criteria.

III. To evaluate progression-free and overall survival after CAR T cell infusion.

IV. To evaluate the time to hematological recovery after CAR T cell infusion. V. To evaluate in vivo CAR T cell expansion and persistence. VI. To evaluate acute GVHD within 6 weeks after infusion of CAR T cells in patients who relapsed after allogeneic hematopoietic cell transplantation (HCT).

VII. To evaluate the incidence of cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS).

EXPLORATORY OBJECTIVES:

I. To evaluate the relationship between cytokine expression and cytokine release syndrome (CRS).

II. To determine predictors of response and mechanisms or resistance to CAR-T cells.

III. To evaluate immune effects by CD83 CAR T cells on peripheral blood T cell subsets, B cells and dendritic cells.

IV. To evaluate the relationship between baseline levels of CD83 expression on AML blasts and response following CAR T cell infusion.

V. To evaluate the relationship between proportion of infused CAR T cell subsets (γδ T cells versus [vs.] αβ T cells) and disease response.

VI. To evaluate immunity after CAR T cell infusion. VII. To determine the rate of successful manufacturing and time required to complete.

VIII. To evaluate for CAR T phenotype, exhaustion, and CAR versus non-CAR subsets associated with response and relapse.

IX. Evaluate the effect of CAR T infusion on quality of life.

OUTLINE:

Patients undergo leukapheresis to obtain peripheral blood mononuclear cells (PBMCs) for CD83 CAR T cell product manufacturing on day -21 and may receive hydroxyurea at the discretion of the treating physician on study. Patients then receive fludarabine intravenously (IV) over 30 minutes and cyclophosphamide IV over 2 hours on days -5 to -3 in the absence of disease progression or unacceptable toxicity. Patients then receive CD83 CAR T cells IV over 15 minutes on day 0. Patients also undergo echocardiography (ECHO) and chest x-ray during screening, blood sample collection throughout the study, and computed tomography (CT) and/or positron emission tomography (PET), as well as lumbar puncture as clinically indicated. In addition, patients may undergo bone marrow aspiration throughout the study.

After completion of study treatment, patients are followed up every 2 weeks for 2 months then at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Karnofsky performance status score ≥ 70%.
* Relapsed or refractory AML based upon ELN 2022 criteria.
* Creatinine clearance: ≥ 40 mL/min (Cockroft-Gault).
* Total bilirubin: ≤ 2mg/dL except for patients with Gilbert's syndrome, hemolysis, or related to disease.
* Aspartate aminotransferase (AST) and alanine transaminase (ALT) < 3.0 x upper limit of normal (ULN).
* Left ventricular (LV) ejection fraction: > 45% and be free of symptomatic congestive heart failure or uncontrolled arrhythmia.
* Oxygen (O2) saturation: ≥ 92% on room air without needs for supplemental O2.
* Absolute lymphocyte count: ≥ 0.2 x 10^9/L, HCT of ≥ 27% and platelets of ≥ 20 x 10^9/L. Transfusion support is allowed to meet HCT and platelet parameters prior to apheresis.
* Life expectancy ≥12 weeks from the time of enrollment, per clinical judgment.
* Negative serum pregnancy test in females of child-bearing potential (FOCBP). FOCBP is defined as any female who has experienced menarche and who has not undergone successful surgical sterilization or who is not postmenopausal.
* If history of allogeneic HCT, must have completed transplant at least 3 months prior, be off immunosuppression, including ruxolitinib, at least 2 weeks prior to apheresis, and have no evidence of GVHD requiring treatment at enrollment.
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and for 12 months following duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Participants must be considered preliminarily eligible for an allogeneic hematopoietic cell transplantation, with potential donors identified per a transplant and cellular therapy consult at Roswell Park Comprehensive Cancer Center.
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* Concomitant systemic glucocorticoid use at a dose equivalent to > 10 mg daily prednisone at the time of apheresis and/or within 4 weeks of CD83 CAR T infusion for any reasons other than GVHD.
* Diagnosis of acute promyelocytic leukemia (APL; AML M3 by French-American-British [FAB] classification).
* Active central nervous system (CNS) leukemia; patients with history of CNS leukemia in complete response (CR) are eligible.
* Patients enrolled in another investigational therapy protocol for their disease within 14 days or 5 half-lives prior to leukapheresis, whichever is shorter.
* Patients requiring agents or any treatments other than hydroxyurea, single agent cytarbine,hypomethylating agents with or without ventoclax and/or targeted agents (i.e., FLT3, IDH2 or IDH1 inhibitors) to control blast counts within 14 days or 5 half-lives (whichever is shorter) prior to lymphodepletion.
* Ongoing uncontrolled serious infection, pulmonary disease or psycho/social concerns.
* HIV seropositivity or active hepatitis B or C infection within (defined by positive polymerase chain reaction [PCR]) 4 weeks of enrollment.
* Other active malignancy within 2 years of study entry, except for basal cell cancer of skin, cervical cancer treated surgically with curative intent or localized prostate cancer managed with observational approach.
* Active grade II-IV acute GVHD in patients with relapsed AML after HCT requiring treatment.
* Prior solid organ transplant.
* Active autoimmune disease requiring immunosuppressive therapy.
* Pregnant or nursing female participants.
* Unwilling or unable to follow protocol requirements.
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) | Up to 28 days
  Will be defined as any adverse events based on Common Terminology Criteria for Adverse Events (CTCAE) version (v)5. Cytokine release syndrome(CRS)/immune effector cell-associated neurotoxicity syndrome will be graded according to American Society for Transplantation and Cellular Therapy (ASTCT) Consensus Guidelines. The DLTs will be summarized by dose level using frequencies and relative frequencies. Will employ the Bayesian optimal interval design to find the maximal tolerated dose (MTD). The target DLT rate for the MTD is = 0.33.

SECONDARY OUTCOMES:
Objective response | At 28 days and 1 year
  Will be determine as the number of patients achieving complete remission, partial remission, and/or morphologic leukemia free state by 2022 European Leukemia Net Response Criteria. Will be summarized by dose level using frequencies and relative frequencies. Rates will be estimated using 95% credible regions obtained by Jeffrey's prior method. As exploratory analyses, comparisons between dose levels may be made using Fisher's exact test.
Overall survival | From treatment initiation until death due to any cause or last follow-up, assessed up to 1 year
  Will be summarized by dose level using cumulative incidence or Kaplan-Meier curves, as appropriate. Estimates of the median times will be obtained with 95% confidence intervals calculated using the log-log transformation. As exploratory analyses, comparisons between dose levels may be made using Gray's or the log-rank test, as appropriate.
Progression-free survival | From treatment initiation until disease progression/relapse, death due to any cause, subsequent treatment (censored), or last follow-up, assessed up to 1 year
  Will be summarized by dose level using cumulative incidence or Kaplan-Meier curves, as appropriate. Estimates of the median times will be obtained with 95% confidence intervals calculated using the log-log transformation. As exploratory analyses, comparisons between dose levels may be made using Gray's or the log-rank test, as appropriate.
Hematologic recovery | At 28 days
  Will be assessed by achieving an absolute neutrophil count recovery (> 0.5 x 10^9/L). Will be summarized by dose level using frequencies and relative frequencies. Rates will be estimated using 95% credible regions obtained by Jeffrey's prior method. As exploratory analyses, comparisons between dose levels may be made using Fisher's exact test.
Time to hematologic recovery | From treatment initiation until hematologic recovery or last follow-up, assessed up to 1 year
  Relapse or death will be considered the competing risk. Will be summarized by dose level using cumulative incidence or Kaplan-Meier curves, as appropriate. Estimates of the median times will be obtained with 95% confidence intervals calculated using the log-log transformation. As exploratory analyses, comparisons between dose levels may be made using Gray's or the log-rank test, as appropriate.
Acute graft-versus-host disease (GVHD) | Up to 6 weeks
  Will be defined as a grade II-IV acute GVHD. Will be summarized by dose level using cumulative incidence or Kaplan-Meier curves, as appropriate. Estimates of the median times will be obtained with 95% confidence intervals calculated using the log-log transformation. As exploratory analyses, comparisons between dose levels may be made using Gray's or the log-rank test, as appropriate.
Time to GVHD | From treatment initiation until grade II-IV GVHD, 6 weeks post infusion, or last follow-up, assessed up to 1 year
  Relapse or death will be considered the competing risk. Will be summarized by dose level using cumulative incidence or Kaplan-Meier curves, as appropriate. Estimates of the median times will be obtained with 95% confidence intervals calculated using the log-log transformation. As exploratory analyses, comparisons between dose levels may be made using Gray's or the log-rank test, as appropriate.
Treatment-related adverse events | Up to 12 months
  Will be defined as by CTCAE v5 and CRS by ASTCT Consensus Grading for CRS and Neurological Toxicity Associated with Immune Effector Cells. Will be summarized by dose level using frequencies and relative frequencies. Rates will be estimated using 95% credible regions obtained by Jeffrey's prior method. As exploratory analyses, comparisons between dose levels may be made using Fisher's exact test.
Time to treatment related adverse event | From treatment initiation until a treatment related adverse event, 12 months post infusion, or last follow-up, assessed up to 1 year
  Relapse or death will be considered the competing risk. Will be summarized by dose level using cumulative incidence or Kaplan-Meier curves, as appropriate. Estimates of the median times will be obtained with 95% confidence intervals calculated using the log-log transformation. As exploratory analyses, comparisons between dose levels may be made using Gray's or the log-rank test, as appropriate
Number of peripheral blood chimeric antigen receptor (CAR) T cells | Up to 1 year
  Will be summarized by dose level and timepoint (pre- and post-therapy) using the mean, median, and standard deviation; and graphically using dot plots. The log absolute number of CD83 CAR T cells per peripheral blood volume will be modeled as a function of dose level, time, their two-way interaction, and a random subject effect using a linear mixed model. Tests about the appropriate contrasts on model estimates will be sued to compare: 1) changes relative to pre-therapy within each dose level, and 2) changes at a given timepoint between dose levels. All model assumptions will be verified graphically, and transformations applied as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Shernan G Holtan, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States